CLINICAL TRIAL: NCT03747640
Title: Self Transcranial Direct Current Stimulation and Mindfulness-based Meditation for Pain in Older Adults With Knee Osteoarthritis (Self tDCS and Meditation for Knee Pain)
Brief Title: Self Transcranial Direct Current Stimulation and Mindfulness-based Meditation for Pain in Older Adults With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Hyochol Ahn, Associate Professor & Theodore J. and Mary E. Trumble Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-SN-18-0885
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- tDCS with mindfulness-based meditation (Experimental): Self Transcranial Direct Current Stimulation (tDCS) with Mindfulness-Based Meditation
  Interventions: Device: Self Transcranial Direct Current Stimulation (tDCS); Behavioral: mindfulness-based meditation
- sham tDCS with sham meditation (Sham Comparator): Sham self Transcranial Direct Current Stimulation (tDCS) with sham Meditation
  Interventions: Device: Sham Self Transcranial Direct Current Stimulation (tDCS); Behavioral: sham meditation

INTERVENTIONS:
Device: Self Transcranial Direct Current Stimulation (tDCS) — tDCS with a constant current intensity of 2 milliamps (mA) will be applied for 20 minutes per session daily for 2 weeks (Monday to Friday) via the Soterix 1x1 tDCS mini-CT Stimulator device (Soterix Medical Inc., New York; 6.5 inches long, 3 inches wide, 0.7 inches thick) with headgear and 5x7 cm saline-soaked surface sponge electrodes.
  Arms: tDCS with mindfulness-based meditation
Behavioral: mindfulness-based meditation — The meditation intervention will be delivered by a recorded device that participants will be given together with the tDCS. All meditation instruction recordings will be done by an experienced mind-body intervention specialist and installed in a user-friendly MP3 player.
  Arms: tDCS with mindfulness-based meditation
Device: Sham Self Transcranial Direct Current Stimulation (tDCS) — For sham stimulation, the electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2 mA current for 30 seconds.
  Arms: sham tDCS with sham meditation
Behavioral: sham meditation — For sham meditation, the participants will be instructed, approximately every 2-3 minutes, to take deep breaths as we sit in meditation. Time spent giving instructions in the sham meditation intervention will be matched to time spent in the mindfulness intervention.
  Arms: sham tDCS with sham meditation

SUMMARY:
The purpose of this study is to determine the feasibility and preliminary efficacy of a two-week self tDCS and mindfulness-based meditation for pain in older adults with knee osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

* self-reported unilateral or bilateral knee OA pain, according to American College of Rheumatology criteria. According to American College of Rheumatology criteria, participants should meet at least 3 of 6 criteria, including age > 50 years, stiffness < 30 minutes, crepitus, bony tenderness, bony enlargement, and no palpable warmth.
* have had knee OA pain in the past 3 months with an average of at least 30 on a 100 Numeric Rating Scale (NRS) for pain
* can speak and read English
* have a device with internet access that can be used for secure video conferencing for real-time remote supervision
* have no plan to change medication regimens for pain throughout the trial
* are able to travel to the coordinating center
* are willing and able to provide written informed consent prior to enrollment

Exclusion Criteria:

* Participants will be excluded if they have concurrent medical conditions that hinder the completion of the protocol, including any of the following
* history of brain surgery, brain tumor, seizure, stroke, or intracranial metal implantation
* serious medical illness, such as uncontrolled hypertension (i.e., systolic blood pressure/ diastolic blood pressure ≥ 150/95 mm Hg), heart failure, or history of acute myocardial infarction
* alcohol/substance abuse
* cognitive impairment
* pregnancy or lactation
* hospitalization within the preceding year for psychiatric illness

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyochol Ahn, PhD, RN, MSN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.47 (6.38) | 59.47 (7.63) | 59.47 (6.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 7 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 2 | 7
  African American | 4 | 4 | 8
  Asian | 5 | 8 | 13
  Hispanic | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Education [Count of Participants; unit: Participants]
  High School' | 2 | 2 | 4
  2-year College | 3 | 1 | 4
  4- year College | 4 | 6 | 10
  Master's Degree | 4 | 2 | 6
  Doctoral Degree | 2 | 4 | 6
Body Mass Index [Mean (Standard Deviation); unit: kg / m^2] | 27.9 (6.35) | 27.17 (5.19) | 27.54 (5.71)
Clinical Pain as Assessed by a Numeric Rating Scale for Pain (NRS) [Mean (Standard Deviation); unit: score on a scale] — The NRS assess average pain over the past 24 hours from 0 (no pain) to 100 (most intense pain imaginable).
  score on a scale | 55.33 (21) | 40.67 (13.35) | 48 (18.83)
Clinical Pain as Assessed by the Western Ontario and McMaster Universities Osteoarthritis Index [Mean (Standard Deviation); unit: score on a scale] — The WOMAC ranges from 0 to 96, with higher scores indicating worse osteoarthritis (O)A pain-related symptoms.
  score on a scale | 42.27 (23.30) | 36.33 (16.14) | 39.30 (19.92)
Experimental Pain Sensitivity as measured by Conditioned Pain Modulation (CPM) [Mean (Standard Deviation); unit: kilograms force (kgf)] — Conditioned Pain Modulation (CPM) was assessed as the change in PPT on the trapezius immediately after the immersion of the contralateral hand up to the wrist in a cold-water bath (Neslab, Portsmouth, NH) at 12 degrees C for one minute. [To assess PPT, a handheld digital pressure algometer (Wagner, Greenwich, CT) was applied at a constant rate of 0.3 kilograms force per centimeter squared (kgf/cm^2) per second to the participant's trapezius. Participants were asked to notify the experimenter when the pressure sensation ''first becomes painful" to assess pressure pain threshold (PPT).]
  kilograms force (kgf) | 0.67 (0.68) | 0.94 (1.25) | .81 (1.00)
Experimental Pain Sensitivity as Assessed by Pressure Pain Threshold, Medial Knee [Mean (Standard Deviation); unit: kilograms force (kgf)] — To assess pressure pain threshold (PPT), a handheld digital pressure algometer (Wagner, Greenwich, CT) was applied at a constant rate of 0.3 kilograms force per centimeter squared (kgf/cm^2) per second to the participant's knee. Participants were asked to notify the experimenter when the pressure sensation ''first becomes painful" to assess pressure pain threshold (PPT).
  kilograms force (kgf) | 3.54 (2.18) | 3.80 (1.56) | 3.67 (1.87)
Experimental Pain Sensitivity as Assessed by Pressure Pain Threshold, lateral Knee [Mean (Standard Deviation); unit: kilograms force (kgf)] — Measure Description: To assess pressure pain threshold (PPT), a handheld digital pressure algometer (Wagner, Greenwich, CT) was applied at a constant rate of 0.3 kilograms force per centimeter squared (kgf/cm^2) per second to the participant's knee. Participants were asked to notify the experimenter when the pressure sensation ''first becomes painful" to assess pressure pain threshold (PPT).
  kilograms force (kgf) | 3.47 (2.18) | 3.96 (1.88) | 3.72 (2.01)
Experimental Pain Sensitivity as Assessed by Cold Pain Intensity [Mean (Standard Deviation); unit: score on a scale] — Participants immersed their hand in a cold water bath, and at thirty seconds after hand immersion, they rated the cold pain intensity on a scale of 0-100. A higher score indicating higher pain intensity
  score on a scale | 78.33 (19.61) | 77.33 (23.14) | 77.83 (21.08)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Pain as Assessed by a Numeric Rating Scale for Pain (NRS)
Description: The NRS assess average pain over the past 24 hours from 0 (no pain) to 100 (most intense pain imaginable).
Time Frame: baseline, 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | -24.67 (12.88) | -3.33 (10.63)

2. Secondary Outcome: Change in Clinical Pain as Assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The WOMAC ranges from 0 to 96, with higher scores indicating worse osteoarthritis (OA) pain-related symptoms.
Time Frame: baseline, 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | -12.60 (17.97) | -0.53 (10.01)

3. Secondary Outcome: Psychosocial Symptoms as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety-short Form
Description: The 7-item PROMIS Anxiety Short Form assesses the pure domain of anxiety in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- tDCS With Mindfulness-based Meditation: Self Transcranial Direct Current Stimulation (tDCS) with Mindfulness-Based Meditation Self Transcranial Direct Current Stimulation (tDCS): tDCS with a constant current intensity of 2 milliamps (mA) will be applied for 20 minutes per session daily for 2 weeks (Monday to Friday) via the Soterix 1x1 tDCS mini-CT Stimulator device (Soterix Medical Inc., New York; 6.5 inches long, 3 inches wide, 0.7 inches thick) with headgear and 5x7 cm saline-soaked surface sponge electrodes.
  mindfulness-based meditation: The meditation intervention will be delivered by a recorded device that participants will be given together with the tDCS. All meditation instruction recordings will be done by an experienced mind-body intervention specialist and installed in a user-friendly MP3 player.
- Sham tDCS With Sham Meditation: Sham self Transcranial Direct Current Stimulation (tDCS) with sham Meditation Sham Self Transcranial Direct Current Stimulation (tDCS): For sham stimulation, the electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2 mA current for 30 seconds.
  sham meditation: For sham meditation, the participants will be instructed, approximately every 2-3 minutes, to take deep breaths as we sit in meditation. Time spent giving instructions in the sham meditation intervention will be matched to time spent in the mindfulness intervention.
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | 17.13 (5.66) | 16.20 (5.41)

4. Secondary Outcome: Psychosocial Symptoms as Assessed by the PROMIS Anxiety-short Form
Description: as for outcome 3
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | 14.27 (6.71) | 14.27 (5.68)

5. Secondary Outcome: Psychosocial Symptoms as Assessed by PROMIS Depression-short Form
Description: The 8-item PROMIS Depression Short Form assesses the pure domain of depression in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | 13.93 (7.74) | 14.00 (5.39)

6. Secondary Outcome: Psychosocial Symptoms as Assessed by PROMIS Depression-short Form
Description: as for outcome 5
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | 11.93 (6.94) | 12.20 (4.83)

7. Secondary Outcome: Psychosocial Symptoms as Assessed by PROMIS Sleep Disturbance-short Form
Description: The 8-item PROMIS Sleep Disturbance Short Form assesses the pure domain of sleep disturbance in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | 23.87 (7.22) | 23.67 (7.49)

8. Secondary Outcome: Psychosocial Symptoms as Assessed by PROMIS Sleep Disturbance-short Form
Description: as for outcome 7
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | 18.27 (4.43) | 21.13 (7.06)

9. Secondary Outcome: Psychosocial Symptoms as Assessed by the Pain Catastrophizing Scale (PCS)
Description: The Pain Catastrophizing Scale (PCS) consists of 13 items assessing three components of catastrophizing: rumination, magnification, and helplessness. Each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time).The PCS total score is computed by summing responses to all 13 items, with total scores ranging from 0 - 52. Higher scores indicate a worse outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | 21.53 (14.46) | 16.73 (13.15)

10. Secondary Outcome: Psychosocial Symptoms as Assessed by the Pain Catastrophizing Scale (PCS)
Description: as for outcome 9
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | 15.80 (13.62) | 14.80 (14.97)

11. Secondary Outcome: Psychosocial Symptoms as Assessed by the Freiburg Mindfulness Inventory (FMI)
Description: The Freiburg Mindfulness Inventory (FMI) is a 14-item instrument. Respondents indicate their experiences relating to the items on a 4-point Likert scale (rarely, occasionally, fairly often and almost always), and the total score is calculated by adding all the scores on the 14 items of the FMI. Total scores range from 14-56, with higher scores indicating higher levels of mindfulness.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | 41.13 (5.60) | 36.40 (7.01)

12. Secondary Outcome: Psychosocial Symptoms as Assessed by the Freiburg Mindfulness Inventory (FMI)
Description: as for outcome 11
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | 42.67 (6.98) | 38.93 (7.43)

13. Secondary Outcome: Change in Experimental Pain Sensitivity as Assessed by Conditioned Pain Modulation
Description: Conditioned Pain Modulation (CPM) was assessed as the change in PPT on the trapezius immediately after the immersion of the contralateral hand up to the wrist in a cold-water bath (Neslab, Portsmouth, NH) at 12 degrees C for one minute. [To assess PPT, a handheld digital pressure algometer (Wagner, Greenwich, CT) was applied at a constant rate of 0.3 kilograms force per centimeter squared (kgf/cm^2) per second to the participant's trapezius. Participants were asked to notify the experimenter when the pressure sensation ''first becomes painful" to assess pressure pain threshold (PPT).]
Time Frame: baseline, 2 weeks
Measure: Mean (Standard Deviation); unit: kilograms force (kgf)
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
kilograms force (kgf) | 0.73 (1.31) | -0.78 (1.17)

14. Secondary Outcome: Number of Participants Who Were Assessed by Functional Near-infrared Spectroscopy (fNIRS)
Description: Pain-related cortical response will be measured using a continuous-wave, multichannel fNIRS imaging system (LIGHTNIRS, Shimadzu, Kyoto, Japan) with three semiconductor lasers at 780, 805, and 830 nm. Optical recordings will be collected during thermal pain stimulation.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
Participants | 15 | 15

15. Secondary Outcome: Number of Participants Who Were Assessed by Functional Near-infrared Spectroscopy
Description: as for outcome 14
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
Participants | 15 | 15

16. Secondary Outcome: Change in Experimental Pain Sensitivity as Assessed by Cold Pain Intensity
Description: Participants immersed their hand in a cold water bath, and at thirty seconds after hand immersion, they rated the cold pain intensity on a scale of 0-100. A higher score indicating higher pain intensity.
Time Frame: baseline, 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
score on a scale | -15.33 (22.40) | 9.67 (19.32)

17. Secondary Outcome: Change in Experimental Pain Sensitivity as Assessed by Pressure Pain Threshold, Lateral Knee
Description: To assess pressure pain threshold (PPT), a handheld digital pressure algometer (Wagner, Greenwich, CT) was applied at a constant rate of 0.3 kilograms force per centimeter squared (kgf/cm^2) per second to the participant's knee. Participants were asked to notify the experimenter when the pressure sensation ''first becomes painful" to assess pressure pain threshold (PPT).
Time Frame: baseline, 2 weeks
Measure: Mean (Standard Deviation); unit: kilograms force (kgf)
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
kilograms force (kgf) | .75 (1.29) | -.71 (0.82)

18. Secondary Outcome: Change in Experimental Pain Sensitivity as Assessed by Pressure Pain Threshold, Medial Knee
Description: as for outcome 17
Time Frame: baseline, 2 weeks
Measure: Mean (Standard Deviation); unit: kilograms force (kgf)
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
Number analyzed (Participants) | 15 | 15
kilograms force (kgf) | .69 (1.16) | -.79 (.58)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | tDCS With Mindfulness-based Meditation | Sham tDCS With Sham Meditation
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03747640/Prot_SAP_000.pdf